CLINICAL TRIAL: NCT05985746
Title: Effectiveness of Augmented Reality in Anatomy Education: The TEACHANATOMY Randomized Clinical Trial
Brief Title: Comparative Study of Augmented Reality vs Traditional Learning in Anatomy Education
Acronym: TEACHANATOMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Lukas Zingg, Doctor of Medicine, Balgrist University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TEACHANATOMY
Record Dates: First submitted 2023-07-17; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Augmented Reality; Anatomy Education
Keywords: Anatomy teaching; Augmented reality; Microsoft HoloLens; Cranial nerves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality (AR) group. (Experimental): - The experimental group will consist of approximately 20 undergraduate medical students. Participants will use the TEACHANATOMY learning application with the HoloLens 2.
  Interventions: Other: Augmented reality group
- Traditional learning (TL) group. (Active Comparator): - The control group will consist of approximately 20 undergraduate medical students. Participants will use traditional learning methods with textbooks, atlases, videos, and online learning programs,
  Interventions: Other: Traditional learning group

INTERVENTIONS:
Other: Augmented reality group — * Study presentation: participants will be given a 10-minute general introduction on the study followed by a 20 minutes tutorial to introduce the HoloLens 2 and the TEACHANATOMY learning platform.
  * Study session: The study session consists of three learning blocks of approximately 20 minutes each, plus a repetition block to assess the acquired knowledge. During the study session participants will be given no time constraints and free breaks.
  * Assessment test: Participants will be assessed with a 30 minutes knowledge assessment test.
  * Final questionnaire: At the end participants will be given a questionnaire to assess adverse health symptoms and user experience.
  Arms: Augmented Reality (AR) group.
Other: Traditional learning group — * Study presentation: participants will be given a 10-minute general introduction on the study followed by a presentation to introduce the study session.
  * Study session: The study session consists of the learning resources most used by students: specific sections from four different neuroanatomy books, access to two websites, two 3D videos, and two online learning programs. During the study session participants will be given no time constraints and free breaks.
  * Assessment test: Participants will be assessed with a 30 minutes knowledge assessment test.
  * Final questionnaire: At the end participants will be given a questionnaire to assess adverse health symptoms and user experience.
  Arms: Traditional learning (TL) group.

SUMMARY:
The goal of this clinical trial is to assess the efficacy of augmented reality (AR) in anatomy teaching.

The main question to answer is: Is 3-Dimensional AR technology more effective than traditional learning methods in anatomy education? In this clinical trial undergraduate medical students with no prior anatomy education will be recruited. Participants in the AR group will learn the anatomy of the cranial nerves with an AR application using Microsoft HoloLens 2, whereas participants in the control group will learn with traditional learning methods (textbooks, atlases, videos, and online learning programs).

DETAILED DESCRIPTION:
Anatomy is a central part in medical training and is traditionally taught through lectures, textbooks, videos and cadaver dissections. Cadaver dissections are important to understand spatial relationships and individual variations of anatomical structures. In many universities, however, financial and ethical considerations, as well as uncommon circumstances such as the COVID-19 pandemic, have restricted access to cadaver dissections. Consequently, new teaching methods based on visual technologies such as augmented reality (AR) are being implemented worldwide. AR can generate realistic 3-dimensional (3D) images overlaid in the real-word environment, merging real and virtual world to provide an interactive learning experience. The use of such technologies in education is still in the early stages, and further research is needed to assess their beneficial impact in knowledge acquisition. The TEACHANATOMY project aim to develop a 3D, interactive AR teaching module focused on the anatomy of the cranial nerves. To assess its potential value in anatomy education, the investigators will perform a study to compare traditional learning methods based on textbooks, videos, and online resources, with the novel AR learning module using the HoloLens 2 (Microsoft Corporation). The goal is to assess whether AR technology can improve anatomical knowledge and enhance student's motivation and engagement.

ELIGIBILITY:
Inclusion Criteria:

* Medical students attending the 1st or 2nd year of undergraduate medical education
* Must not have prior neuroanatomical education

Exclusion Criteria:

* Epilepsy
* Binocular vision disorder such as strabismus
* Current head and/or neck injuries
* Inflammation of the scalp and/or eye
* Amputations or partial amputations of the hands

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-21 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Knowledge acquisition | Immediately after the study session, Day 1
  The primary outcome will consist of the score in the final theoretical and practical tests. The theoretical test consist of 23 single and multiple-choice questions in which participants will be required to recognize and name the 12 cranial nerves, differentiate their main functions and the typology (sensory, motor, mixed), explain the relationships between their structure and function, and recognize lesions using case studies. In the practical part, participants will be required to mark specific nerves in a 3D-printed anatomical skull model. The duration of the test will be of 30 minutes.

SECONDARY OUTCOMES:
Adverse Health Symptoms | Immediately after the knowledge acquisition test, Day 1.
  Secondary outcomes will include adverse health symptoms, evaluated with a questionnaire to assess presence and severity of general symptoms (General discomfort, Fatigue, Headache, Dizziness, Nausea, Concentration problems, Disorientation, Neck stiffness/neck pain, No symptoms) and eye-related symptoms (Blurred vision, Difficulty focusing, Double-vision, Dry eyes No symptoms). Presence and severity of symptoms will be rated on a Likert scale from 1 (almost imperceptible) to 10 (extreme).
User experience | Immediately after the knowledge acquisition test, Day 1.
  User experience will be assessed using an adapted NASA Task Load Index (5 questions, range, 1-10, with lower scores indicating lower cognitive workload) plus additional 10-point Likert scale and open-ended questions, in which participants were asked to rank their comfort with the material and hardware and the teaching effectiveness of the software or of the traditional learning methods to learn the anatomy of the cranial nerves

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Zingg, Cand. Med., Principal Investigator — Balgrust University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Z, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moro C, Stromberga Z, Raikos A, Stirling A. The effectiveness of virtual and augmented reality in health sciences and medical anatomy. Anat Sci Educ. 2017 Nov;10(6):549-559. doi: 10.1002/ase.1696. Epub 2017 Apr 17. PMID 28419750
- [Background] Bolek KA, De Jong G, Henssen D. The effectiveness of the use of augmented reality in anatomy education: a systematic review and meta-analysis. Sci Rep. 2021 Jul 27;11(1):15292. doi: 10.1038/s41598-021-94721-4. PMID 34315955
- [Background] Chytas D, Johnson EO, Piagkou M, Mazarakis A, Babis GC, Chronopoulos E, Nikolaou VS, Lazaridis N, Natsis K. The role of augmented reality in Anatomical education: An overview. Ann Anat. 2020 May;229:151463. doi: 10.1016/j.aanat.2020.151463. Epub 2020 Jan 21. PMID 31978568
- [Background] Curran VR, Xu X, Aydin MY, Meruvia-Pastor O. Use of Extended Reality in Medical Education: An Integrative Review. Med Sci Educ. 2022 Dec 19;33(1):275-286. doi: 10.1007/s40670-022-01698-4. eCollection 2023 Feb. PMID 36569366
- [Background] Gsaxner C, Li J, Pepe A, Jin Y, Kleesiek J, Schmalstieg D, Egger J. The HoloLens in medicine: A systematic review and taxonomy. Med Image Anal. 2023 Apr;85:102757. doi: 10.1016/j.media.2023.102757. Epub 2023 Jan 21. PMID 36706637
- [Background] McBain KA, Habib R, Laggis G, Quaiattini A, M Ventura N, Noel GPJC. Scoping review: The use of augmented reality in clinical anatomical education and its assessment tools. Anat Sci Educ. 2022 Jul;15(4):765-796. doi: 10.1002/ase.2155. Epub 2022 Jan 19. PMID 34800073
- [Background] Moro C, Birt J, Stromberga Z, Phelps C, Clark J, Glasziou P, Scott AM. Virtual and Augmented Reality Enhancements to Medical and Science Student Physiology and Anatomy Test Performance: A Systematic Review and Meta-Analysis. Anat Sci Educ. 2021 May;14(3):368-376. doi: 10.1002/ase.2049. Epub 2021 Feb 26. PMID 33378557
- [Background] Navab N, Martin-Gomez A, Seibold M, Sommersperger M, Song T, Winkler A, Yu K, Eck U. Medical Augmented Reality: Definition, Principle Components, Domain Modeling, and Design-Development-Validation Process. J Imaging. 2022 Dec 23;9(1):4. doi: 10.3390/jimaging9010004. PMID 36662102
- [Background] Stojanovska M, Tingle G, Tan L, Ulrey L, Simonson-Shick S, Mlakar J, Eastman H, Gotschall R, Boscia A, Enterline R, Henninger E, Herrmann KA, Simpson SW, Griswold MA, Wish-Baratz S. Mixed Reality Anatomy Using Microsoft HoloLens and Cadaveric Dissection: A Comparative Effectiveness Study. Med Sci Educ. 2019 Nov 15;30(1):173-178. doi: 10.1007/s40670-019-00834-x. eCollection 2020 Mar. PMID 34457656
- [Background] Stromberga Z, Phelps C, Smith J, Moro C. Teaching with Disruptive Technology: The Use of Augmented, Virtual, and Mixed Reality (HoloLens) for Disease Education. Adv Exp Med Biol. 2021;1317:147-162. doi: 10.1007/978-3-030-61125-5_8. PMID 33945136
- [Background] Uruthiralingam U, Rea PM. Augmented and Virtual Reality in Anatomical Education - A Systematic Review. Adv Exp Med Biol. 2020;1235:89-101. doi: 10.1007/978-3-030-37639-0_5. PMID 32488637
- [Background] Ghosh SK. Cadaveric dissection as an educational tool for anatomical sciences in the 21st century. Anat Sci Educ. 2017 Jun;10(3):286-299. doi: 10.1002/ase.1649. Epub 2016 Aug 30. PMID 27574911
- See also: Microsoft HoloLens 2 device — https://www.microsoft.com/en-us/hololens/hardware#document-experiences